CLINICAL TRIAL: NCT03008785
Title: Effect of Isoflavone Supplementation Associated With Physical Exercise on Blood Pressure, Lipic and Inflamatory Profile, Body Composition and Hydratation and Climacteric Symptoms in Postmenopausal Women
Brief Title: Effect of Isoflavone Supplementation Associated With Physical Exercise in the Health Parameters of Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Juliene Gonçalves Costa, Guilherme Morais Puga PhD, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE: 40622414.9.0000.5152
Record Dates: First submitted 2016-12-28; First posted 2017-01-02 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Bloodpressure
Keywords: isoflavone; blood pressure; climateric symptoms; exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Isoflavones

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- group isoflavone and exercise (Experimental): The isoflavone group received daily 100mg of isoflavones.
  Interventions: Other: exercise; Other: isoflavone
- group placebo and exercise (Experimental): The placebo group received 100mg containing starch of corn.
  Interventions: Other: exercise; Other: Placebo

INTERVENTIONS:
Other: exercise — The training program consisted of aerobic and resisted combined physical exercises performed during 10 weeks, three times weekly with 45 minutes sessions: 5 minutes of warm-up on treadmill, 20 minutes of aerobic exercises and 20 minutes of resistance exercises.
Other: isoflavone — Daily supplementation in 1 capsule per day of 100mg of isoflavones (containing 3.3% genistein, 93.5% dadzein and 3.2% glycitein).
  Arms: group isoflavone and exercise
Other: Placebo — Daily supplementation in 1 capsule per day containing starch of corn.
  Arms: group placebo and exercise

SUMMARY:
This study evaluate if 10 weeks of mixed exercise combined with isoflavones could have greater effects on climacteric symptoms, body composition and hydratation, lipidic and inflamatory profile than exercise alone in postmenopausal women. the participants will be randomly assigned to the group: placebo and exercise or 100mg of isoflavone and exercise.

DETAILED DESCRIPTION:
Several endocrine metabolic changes occur during the climacteric period, due to the lack of estrogen and also by the aging process and some studies show that ingestion of isoflavones by postmenopausal women may have benefits. Theoretically the isoflavone potentiate the effects obtained during exercise

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal woman
* to be able to practice exercises on treadmill and weight exercises
* without physical complications that prevent the execution of physical exercises
* have no history of cardiovascular disease, diabetes, renal pathologies or hypertension

Exclusion Criteria:

* smokers
* use hormone therapy or isoflavone
* use drugs that interfere with lipid and antihypertensive metabolism

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-02; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | Change in blood pressure in 10 weeks intervention
  Evaluate change in blood pressure through ambulatory 24-hour blood pressure monitoring used before the begin of intervention and after 10 weeks.

SECONDARY OUTCOMES:
Climateric Symptoms (Kupperman-Blatt Index) | before and after 10 weeks
  Evaluate the intensity of climateric symptoms using the Kupperman-Blatt Index questionnaire. Consists of 11 questions in which the symptoms are given numerical values according to their intensity .
Climateric Symptoms (Cervantes Scale) | before the begin the intervention and after 10 weeks
  Evaluate the intensity of climateric symptoms using the Cervantes Scale questionnaire. Composed of 31 questions distributed in four domains and 6 possibilities of answer.
Climateric Symptoms (Menopause Rating Scale) | before and after 10 weeks
  Evaluate the intensity of climateric symptoms using the Menopause Rating Scale questionnaire. Composed of eleven questions, with five possible answers, Symptoms divided into somatovegetative, psychological and urogenital domains may be classified as absent, mild, moderate, severe and very severe. With a general score ranging from 0 to 55 points
Lipid profile (enzymatic colorimetric method) | before and after 10 weeks
  The concentrations in mg/dL of total cholesterol, triglycerides, HDL cholesterol, LDL cholesterol and uric acid will be made through the enzymatic colorimetric method. The glucose will be analyzed by the enzymatic method and the glycated hemoglobin A1c by the turbidimetry method.
Human cytokines (Flow Cytometry) | before and after 10 weeks
  Measurement in pg/mL of the production of human cytokines (IL-8, IL-1β, IL-6, TNF ( tumor necrosis factor), IL-10 and IL-12p70) in serum samples will be performed by the flow cytometry (FACSCantoII BDTM) Human Inflammatory Cytokines Kit "(BD ™ Cytometric Bead Array (CBA), BD Biosciences, San Jose, CA, USA) according to the manufacturer's instructions.
Antioxidant capacity | before and after 10 weeks
  The total antioxidant capacity will be evaluated in plasma and saliva using the FRAP (Ferric-Absorbing Ability of Plasma) methodology (Benzie and Strain, 1999).
Total protein | before and after 10 weeks
  The determination of the total salivary and plasma protein will be performed by the Bradfort method (Bradford, 1976) adapted for microplate
Body Composition | before and after 10 weeks
  Bioelectrical impedance (Biodynamics, model 450c, EUA) will be used to determine absolute and relative extracellular mass and body cell mass.
Phase Angle | before and after 10 weeks
  Phase angle in degrees (o) was calculated using the equation (Reactance/Resistance)
  *(180/л) using a values obtained on bioelectrical impedance (Biodynamics, model 450c, EUA)
Oxidative stress (SOD, Catalase and TBARS activity) | before and after 10 weeks
  The enzyme superoxide dismutase (SOD) will be dosed from the auto oxidation capacity of pyrogallol, a process dependent on the superoxide radical (Fernandes et al., 2011). . Catalase activity in saliva will be determined based on the decrease in absorbance of hydrogen peroxide (H2O2) (Aebi, 1984). Thiobarbituric acid reactive substances (TBARS) will be detected by the Yagi method (Yagi, 1998).

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Puga, PhD, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Guilherme Morais Puga, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Acharjee S, Zhou JR, Elajami TK, Welty FK. Effect of soy nuts and equol status on blood pressure, lipids and inflammation in postmenopausal women stratified by metabolic syndrome status. Metabolism. 2015 Feb;64(2):236-43. doi: 10.1016/j.metabol.2014.09.005. Epub 2014 Oct 5. PMID 25441251
- [Result] Lebon J, Riesco E, Tessier D, Dionne IJ. Additive effects of isoflavones and exercise training on inflammatory cytokines and body composition in overweight and obese postmenopausal women: a randomized controlled trial. Menopause. 2014 Aug;21(8):869-75. doi: 10.1097/GME.0000000000000177. PMID 24378766
- [Derived] Barbosa CD, Costa JG, Giolo JS, Rossato LT, Nahas PC, Mariano IM, Batista JP, Puga GM, de Oliveira EP. Isoflavone supplementation plus combined aerobic and resistance exercise do not change phase angle values in postmenopausal women: A randomized placebo-controlled clinical trial. Exp Gerontol. 2019 Mar;117:31-37. doi: 10.1016/j.exger.2018.08.007. Epub 2018 Sep 1. PMID 30176281